CLINICAL TRIAL: NCT02257658
Title: Doxycycline Prophylaxis or Incentive Payments to Reduce Incident Syphilis Among HIV- Infected Men Who Have Sex With Men Who Continue to Engage in High Risk Sex: A Randomized, Controlled Pilot Study
Brief Title: Efficacy of Doxycycline Prophylaxis to Reduce Syphilis in High-Risk, HIV-Positive MSM
Acronym: DPMSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Los Angeles LGBT Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Matthew Beymer, Epidemiologist, Health and Mental Health Services, Los Angeles LGBT Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHS 398/2590
Record Dates: First submitted 2014-10-01; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Syphilis
Keywords: Men who have Sex with Men; HIV-positive; Syphilis; Contingency Management
MeSH Terms: conditions — Syphilis; Homosexuality; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Experimental): Subjects in the doxycycyline arm will receive Doxycycline, oral, 100 mg, once daily for 36 weeks.
  Interventions: Drug: Doxycycyline
- Incentive (Active Comparator): Subjects in the incentive arm will receive escalating payments for remaining STI free at Weeks 12, 24 and 36.
  Interventions: Behavioral: Incentive

INTERVENTIONS:
Drug: Doxycycyline
  Arms: Doxycycline
Behavioral: Incentive
  Arms: Incentive

SUMMARY:
This pilot study will investigate the feasibility of conducting a large, randomized trial comparing a structural intervention to contingency management to reduce incident syphilis infections in an especially high risk group: HIV+ men who have sex with men (MSM) who have had syphilis twice or more since their HIV diagnosis. Subjects will be randomized to receive either QD doxycycline as syphilis prophylaxis or a financial incentive to remain STI free. The investigators will : 1) measure adherence to study visits in both arms; 2) measure adherence to the prophylaxis regimen; 3) measure any changes in risk behaviors among study participants and 4) to the extent possible in a small pilot study of short duration, compare effectiveness of doxycycline with that of a monetary incentive for remaining STI free.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected MSM or transgender women who have sex with men
* At least two documented and adequately treated episodes of syphilis since HIV diagnosis

Exclusion Criteria:

* Had a known allergy or intolerance to doxycycline
* Abused alcohol or other substances which in the opinion of the investigators would jeopardize adherence to study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Measure changes in the incidence of Syphilis, Gonorrhea and Chlamydia at 12 weeks, 24 weeks, 26 weeks and 48 weeks in the Doxycycline Arm and Contingency Management Arms | 12 Weeks, 24 Weeks, 36 Weeks and 48 Weeks

SECONDARY OUTCOMES:
Measure adherence to study visits in the Doxycycline and Contingency Management Arms at Weeks 12, 24, 36 and 48 | 12 Weeks, 24 Weeks, 36 Weeks and 48 Weeks
Measure adherence to daily Doxycycline Use using Blood Samples in the Doxycycline Arm at Weeks 12, 24 and 36 | 12 Weeks, 24 Weeks and 36 Weeks
  At Weeks 12, 24 and 36, blood samples were drawn from participants in the Doxycycline arm and sent to a lab to measure doxycyline levels in each participant in the Doxycyline Arm. The purpose of this outcome is to determine if individuals in the Doxycycline Arm are consistently adhering to the daily regimen of the drug.
Measure changes in self-report sexual risk behaviors (e.g., condom use, drug use and number of partners) in the Doxycycline and Contingency Management Arms at Weeks 12, 24 and 36 | 12 Weeks, 24 Weeks and 36 Weeks
  Prior to having labs drawn, participants in both the Doxycycline and Contingency Management Arms were asked about their risk behaviors in the past three months including: meth use, condom use with casual partners, condom use with regular partners, condom use with a main partner, number of casual sexual partners and number of regular sexual partners.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Klausner, MD, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Background] Celum CL. Sexually transmitted infections and HIV: epidemiology and interventions. Top HIV Med. 2010 Oct-Nov;18(4):138-42. PMID 21107013
- [Background] Goh BT. Syphilis in adults. Sex Transm Infect. 2005 Dec;81(6):448-52. doi: 10.1136/sti.2005.015875. PMID 16326843
- [Background] Lynn WA, Lightman S. Syphilis and HIV: a dangerous combination. Lancet Infect Dis. 2004 Jul;4(7):456-66. doi: 10.1016/S1473-3099(04)01061-8. PMID 15219556
- [Background] Centers for Disease Control and Prevention (CDC). Outbreak of syphilis among men who have sex with men--Southern California, 2000. MMWR Morb Mortal Wkly Rep. 2001 Feb 23;50(7):117-20. PMID 11393490
- [Background] Horberg MA, Ranatunga DK, Quesenberry CP, Klein DB, Silverberg MJ. Syphilis epidemiology and clinical outcomes in HIV-infected and HIV-uninfected patients in Kaiser Permanente Northern California. Sex Transm Dis. 2010 Jan;37(1):53-8. doi: 10.1097/OLQ.0b013e3181b6f0cc. PMID 19734820
- [Background] Marcus JL, Katz KA, Bernstein KT, Nieri G, Philip SS. Syphilis testing behavior following diagnosis with early syphilis among men who have sex with men--San Francisco, 2005-2008. Sex Transm Dis. 2011 Jan;38(1):24-9. doi: 10.1097/OLQ.0b013e3181ea170b. PMID 20679965
- [Background] Fleming DT, Wasserheit JN. From epidemiological synergy to public health policy and practice: the contribution of other sexually transmitted diseases to sexual transmission of HIV infection. Sex Transm Infect. 1999 Feb;75(1):3-17. doi: 10.1136/sti.75.1.3. PMID 10448335